CLINICAL TRIAL: NCT05902806
Title: Evaluation of the Gastro-intestinal Tolerance, Nutritional Intake, and Acceptability of an Upgraded Composition of an Enteral Tube Feed for Adults in Need of Long Term Nutritional Support (Peacock Butterfly)
Brief Title: Evaluation of the Gastro-intestinal Tolerance of an Upgraded Composition of an Enteral Tube Feed for Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SBB22R&56358
Record Dates: First submitted 2023-04-21; First posted 2023-06-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Enteral Tube Nutrition

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, multi-centre, multi-country, exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of current tube feed to intervention feed with upgraded composition (Experimental): Subjects will use their own current practice tube feed for 1 week (baseline period) and will switch to the intervention tube feed with an upgraded composition with a comparable energy density and fiber content as their current tube for 2 weeks (intervention period). Since four different products will be evaluated (product A-D), there will be 4 study groups
  Interventions: Dietary Supplement: Upgraded tube feed

INTERVENTIONS:
Dietary Supplement: Upgraded tube feed — Total duration of study: 4 weeks; 1 week on current tube feed followed by 2 weeks on upgraded tube feed comparable in energy density and fiber content as their current tube feed. The tube feeding regimen is similar to pre study feeding regimen. There will then be a one week follow up period.

SUMMARY:
This study evaluates the gastro-intestinal tolerance, nutritional intake, and acceptability of an upgraded composition of an enteral tube feed for adults in need of long term nutritional support.

DETAILED DESCRIPTION:
Four current tube feed products are upgraded with the same product composition and will be investigated in this study. Subjects will be asked to continue with their current tube feeding for 7 days (baseline period) and asked to complete a daily gastro-intestinal tolerance questionnaire. On Day 8, the subjects will switch to one of four upgraded tube feeding products for 14 days (intervention period). The subjects are asked to complete the same gastro-intestinal tolerance questionnaire for again 7 days. On Day 21 (end of intervention), the subjects will return to their original tube feed product and the investigator will follow up on how they are feeling to evaluate tolerability and product acceptability.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Using either an enteral tube feed with approximately 1.0 or 1.5 kcal/mL with or without fibers via a nasogastric tube (NGT), nasojejunal (NJT) or Percutaneous Endoscopic Gastrostomy (PEG) for at least 4 weeks prior to screening
3. Actual and expected average daily intake of enteral nutrition at least 1000 kcal for at least 21 days after the start of baseline period
4. Written informed consent from subject (or impartial witness after verbal consent of subject)

Exclusion Criteria:

1. Subjects receiving total parental feeding (TPN) 2. Gastro-intestinal surgery or any other surgery involving general anaesthesia within 2 weeks prior to screening 3. Subjects with major hepatic or renal dysfunction in the opinion of the Investigator 4. Subjects currently in the intensive care unit 5. Active/flare up condition of chronic illnesses in small or large intestines in the opinion of the Investigator (e.g., active inflammation/flare up of Crohn's disease or ulcerative colitis) within 2 weeks prior to screening, 6. Subjects experiencing cancer treatment-related diarrhea within 2 weeks prior to screening 7. Presence of colostomy or other faecal diversion 8. Known intolerance or allergy to ingredients of study product (e.g. galactosemia, allergy to soy) 9. Inability of the subject to answer the study diary or questionnaires due to e.g., being unconscious, cognitive impairment, or dementia, in the opinion of the Investigator 10. Known pregnancy or lactation 11. Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements 12. Active participation in any other clinical study involving investigational or marketed products concomitantly or within four weeks prior to entry into the study in the opinion of the Investigator

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Gastro-intestinal tolerance | 7 days in the 1-week baseline period
  self-reported GI symptoms with a GI symptom questionnaire
Gastro-intestinal tolerance | 7 days in the second week of the 2-week intervention period
  self-reported GI symptoms with a GI symptom questionnaire
bowel movement pattern | 7 days in the 1-week baseline period
  Self reported bowel movement pattern with the 7-point Bristol Stool Form Scale (BSFS) ranging from "1" (indicating separate, hard lumps) to "7", which stands for entirely liquid, watery stool without any hard components
bowel movement pattern | 7 days in the second week of the 2-week intervention period
  Self reported bowel movement pattern with the 7-point Bristol Stool Form Scale (BSFS) ranging from "1" (indicating separate, hard lumps) to "7", which stands for entirely liquid, watery stool without any hard components

SECONDARY OUTCOMES:
Volume of tube feed administration | 7 days in the 1-week baseline period, 7 days in the first week of the 2-week intervention period, and 7 days in the second week of the 2-week intervention period (i.e., on a daily basis during the entire study duration).
  Self reported volume of feed administered
Difference between prescribed volume of tube feed administration by Health Care Professional and actual daily self-reported administrated volume of tube feed | 7 days in the 1-week baseline period, 7 days in the first week of the 2-week intervention period, and 7 days in the second week of the 2-week intervention period (i.e., on a daily basis during the entire study duration).
  Product compliance
Use of complementary feeding with a questionnaire ((use of normal foods, oral nutritional supplements, parenteral feeding: Yes/No) | 7 days in the 1-week baseline period, 7 days in the first week of the 2-week intervention period, and 7 days in the second week of the 2-week intervention period (i.e., on a daily basis during the entire study duration).
  Self reported complementary feeding
Product acceptability with a questionnaire | Day 7 end of baseline period regarding the current tube feed
  Self reported product acceptability
Product acceptability with a questionnaire | Day 21 (end of intervention period regarding the upgraded tube feed)
  Self reported product acceptability
Anthropometrics | Baseline Day 1
  Body Height (cm)
Anthropometrics | Baseline Day 1
  Body weight (kg)
Anthropometrics | Baseline Day 7
  Body weight (kg)
Anthropometrics | Intervention Day 7
  Body weight (kg)
Anthropometrics | Intervention Day 14
  Body weight (kg)
Anthropometrics | Intervention Day 21
  Body weight (kg)
Anthropometrics | Baseline Day 1
  Body mass index (kg/m^2)
Anthropometrics | Baseline Day 7
  Body mass index (kg/m^2)
Anthropometrics | Intervention Day 7
  Body mass index (kg/m^2)
Anthropometrics | Intervention Day 14
  Body mass index (kg/m^2)
Anthropometrics | Intervention Day 21
  Body mass index (kg/m^2)

OTHER OUTCOMES:
Medication | 7 days in the 1-week baseline period, 7 days in the first week of the 2-week intervention period, and 7 days in the second week of the 2-week intervention period (i.e., on a daily basis during the entire study duration
  Self reported use of predefined relevant medication with questionnaire (e.g. GI related medication like use of laxatives, antidiarrheals)

CONTACTS AND LOCATIONS:
Locations (1):
- QClinical, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No